CLINICAL TRIAL: NCT07210320
Title: An Open-label, Two-Part, Partially Randomized Single-Dose Crossover Study Evaluating the Safety, Tolerability, and Pharmacokinetics of L-dipivefrin (IN-001) Sublingual Spray in Comparison to Epinephrine 0.3 mg Manual Intramuscular Injection and Epinephrine 0.3 mg Auto-injection in Healthy Adult Volunteers Under Fasted Conditions
Brief Title: PK/PD Study of IN-001 Sublingual Spray in Healthy Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Insignis Therapeutics, Inc. (Industry)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ITI-25-001
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Food Allergy; Anaphylaxis; Food Hypersensitivity; Food Allergy Peanut
Keywords: Type 1 allergy, epinephrine, anaphylaxis, food allergy
MeSH Terms: conditions — Food Hypersensitivity; Anaphylaxis; Peanut Hypersensitivity | interventions — Epinephrine; Needles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment Period 1 (Active Comparator): EpiPen 0.3 mg
  Interventions: Drug: Epinephrine Auto-Injector 0.3 mg/0.3 mL
- Treatment Period 2 (Active Comparator): Epinephrine 0.3 mg IM
  Interventions: Drug: Epinephrine 0.3 mg intramuscular manual injection via a syringe and needle
- Treatment Period 3 (Experimental): IN-001 Sublingual Spray
  Interventions: Drug: IN-001 9.06 mg Sublingual Spray
- Treatment Period 4 (Experimental): IN-001 Sublingual Spray
  Interventions: Drug: IN-001 13.59 mg Sublingual Spray

INTERVENTIONS:
Drug: Epinephrine Auto-Injector 0.3 mg/0.3 mL — Epinephrine injection
  Other Names: Epipen
  Arms: Treatment Period 1
Drug: Epinephrine 0.3 mg intramuscular manual injection via a syringe and needle — Epinephrine injection
  Other Names: Adrenalin
  Arms: Treatment Period 2
Drug: IN-001 9.06 mg Sublingual Spray — Sublingual Spray
  Other Names: IN-001
  Arms: Treatment Period 3
Drug: IN-001 13.59 mg Sublingual Spray — Sublingual Spray
  Other Names: IN-001
  Arms: Treatment Period 4

SUMMARY:
This is an open-label, two-part study to assess the pharmacokinetics (PK) and pharmacodynamics (PD) of epinephrine administered as a single dose of L-dipivefrin (IN-001) sublingual spray in healthy adults. For both parts of the study, participants will undergo at least 10 hours of fasting prior to dosing. Part 1 of the study focuses on IN-001 dose/formulation exploration in a small number of participants (N=6) to help select the most appropriate dose/formulation to be used in Part 2 of the study in a larger number of participants (N=24).

DETAILED DESCRIPTION:
This is an open-label, two-part, partially randomized single-dose crossover study to assess the pharmacokinetics (PK) and pharmacodynamics (PD) of epinephrine administered as a single dose of L-dipivefrin (IN-001) sublingual spray in healthy adults.

Part 1 of the study will have four Treatment Periods testing two doses of IN-001 Sublingual Spray (Test Products) and two doses of approved epinephrine injection products (Reference Products). All participants will receive the same study drug and dose within each of the four Treatment Periods. There will be no randomization in Part 1 of the study. In Period 1, all participants will receive a single dose of EpiPen® (Epinephrine Injection) Auto-Injector 0.3 mg/0.3 mL of Mylan Specialty L.P., USA, once, in the morning after at least 10 hours of fasting. In Period 2, all participants will receive a single dose of Epinephrine 0.3 mg intramuscular manual injection via a syringe and needle, once, in the morning after at least 10 hours of fasting. In Period 3, all participants will receive a single dose of L-dipivefrin (IN-001) 9.06 mg Sublingual Spray of Insignis Therapeutics, Inc., in the morning after at least 10 hours of fasting. In Period 4, all participants will receive a single dose of L-dipivefrin (IN-001) 13.59 mg Sublingual Spray of Insignis Therapeutics, Inc., in the morning after at least 10 hours of pasting. Following Periods 1 and 2, a washout period of at least 24 hours will be observed. Following Period 3, a washout period of 7 days will be observed before Period 4 dosing. Safety and tolerability will be assessed throughout the study.

Part 2 of this study is an open-label, three-period, randomized single-dose study. Participants will be randomized in a 1:1:1 allocation to determine the sequence in which they will be assigned to receive the study medications in Periods 1, 2, and 3. During each period, participants will receive a single dose of one of the three study products. By the end of the study, each participant will have received all three products through a crossover design. The following are the allocations to which participants will be randomized:

* The selected dose from Part 1 of either L-dipivefrin (IN-001) 9.06 mg or 13.59 mg Sublingual Spray by Insignis Therapeutics, Inc., once, in the morning after at least 10 hours of fasting.
* EpiPen® (Epinephrine Injection) Auto-Injector 0.3 mg/0.3 mL of Mylan Specialty L.P., USA, once, in the morning after at least 10 hours of fasting.
* Epinephrine 0.3 mg intramuscular injection, once, in the morning after at least 10 hours of fasting.

Following Periods 1 and 2, there will be a washout period of at least 24 hours that will be observed. Safety and tolerability will be assessed throughout the study.

Participants will exit the study after treatment Period 3 following completion of the 6-hour safety assessments and a 24-hour post-dose follow-up phone call. In the event that a participant completes the trial with a laboratory abnormality or unresolved adverse event (AE), the Investigator will attempt to provide follow-up until a satisfactory clinical resolution of the AE or laboratory result is achieved.

Up to 30 participants are planned to be enrolled in the trial overall. Up to six participants will be dosed Part 1 and up to 24 participants will be dosed in Part 2.

ELIGIBILITY:
Inclusion Criteria:

* To participate in this trial, volunteers must meet all of the inclusion criteria listed below:

  1. Age > 18 years of age and < 45 years of age.
  2. Women of childbearing potential or men with childbearing potential partners must agree that the participant and/or their partner will use the following effective methods of birth control from screening visit until 14 days after the last dose of study drug:

     1. Abstinence
     2. Hormonal contraceptives for at least one month prior to Screening
     3. Double barrier (e.g., diaphragm with spermicide, condom with spermicide)
     4. Intrauterine device (IUD)
     5. Surgically sterile (e.g., bilateral tubal ligation, total or partial hysterectomy, or bilateral oophorectomy)

        * Note: Females will be considered post-menopausal if they

          * are at least 45 years of age with amenorrhea for at least one year, or
          * received bilateral oophorectomy with or without a hysterectomy.
  3. BMI > 18.50 and < 29.90 kg/m2 (using formula BMI = weight (kg)/height (m2).
  4. All clinical laboratory test results (e.g., hematology, chemistry, urinalysis) are within normal limits or considered not clinically significant by Investigator.
  5. Serum pseudocholinesterase activity is within normal limits or considered not clinically significant by Investigator.
  6. Physical examination (excluding genital and rectal exams) is normal or considered not clinically significant by Investigator.
  7. Vital signs measurements (pulse rate, blood pressure, temperature, and respiratory rate) are normal or considered not clinically significant by Investigator, while seated or semi-recumbent and after 5 minutes of rest. Normal vital sign ranges are listed below:

     1. Systolic blood pressure: 90 - 140 mmHg
     2. Diastolic blood pressure: 50 - 90 mmHg
     3. Pulse rate: 45 - 100 beats per minute (bpm)
     4. Oral body temperature: 35.0°C - 37.5°C
  8. 12-lead electrocardiogram (ECG) is normal or considered not clinically significant by Investigator.
  9. Participants must agree to not consume caffeine and/or xanthine containing products (i.e., coffee, tea, chocolate, caffeine-containing sodas, etc.), grapefruit and grapefruit containing products, and poppyseed containing foods within 48 hours prior to Period 1 check-in.
  10. Able to comply with study procedures, in the opinion of the Investigator(s).
  11. Willing to provide written consent for screening procedures. Legally authorized representatives will not be allowed to sign on behalf of participants in this trial.

Exclusion Criteria:

* To participate in this trial, volunteers must not meet any of the exclusion criteria listed below:

  1. Resident of a care facility, incarcerated individual, or individual in residential treatment facilities.
  2. Pregnant and/or breastfeeding.

     1. Females of childbearing potential should have a negative pregnancy test.
     2. Females must agree to refrain from breastfeeding from screening visit through 14 days after the last dose of study drug.
  3. Known history of Human Immunodeficiency Virus (HIV) 1 & 2 and hepatitis B & C virus.
  4. Clinically significant history of alcoholism within the last 12 months, per Investigator's discretion. Participants must

     a. have a negative breath alcohol test at screening. b. agree to abstain from using alcohol for 7 days prior to dosing in Period 1 until the end of study.
  5. Clinically significant history of addiction, abuse, and misuse of any drug, per the Investigator's discretion. Participants must

     a. have a negative drug test for substances of abuse at screening. b. agree to abstain from using drugs for 7 days prior to dosing in Period 1 until the end of study.
  6. Use of tobacco/nicotine containing products (e.g., chewing tobacco, smoking cigarettes, and/or electronic cigarettes) within the last 12 months. Participants must agree to abstain from using tobacco/nicotine containing products from the screening visit until the end of study.
  7. Use of or planned use of any investigational products (i.e., dosing in any clinical investigation) within 30 days prior to Period 1 dosing or within 10 half-lives of the investigational agent previously taken (whichever is longer).
  8. Use of or planned use of any prescription medications, except hormonal contraceptives, within 14 days prior to Period 1 dosing.
  9. Use of or planned use of any over-the-counter medications (e.g., aspirin, ibuprofen, antacids, etc.) within 5 days prior to Period 1 dosing.
  10. Use of or planned use of hormone replacement therapy within 90 days prior to Period 1 dosing.
  11. Use of or planned use of any of the following medications within 30 days prior to Period 1 dosing:

      1. Ergot alkaloids
      2. Cardiac glycosides
      3. Diuretics
      4. Anti-arrhythmic medications
      5. Tricyclic antidepressants
      6. Monoamine oxidase inhibitors
      7. Levothyroxine sodium
      8. Antihistamines, including chlorpheniramine and diphenhydramine
      9. Tripelennamine
      10. Propranolol
      11. Phentolamine
      12. Proton pump inhibitors
      13. Antihypertensives
      14. Chlorpromazine
      15. Ethosuximide
      16. Haloperidol
      17. Lithium carbonate
      18. Meperidine
      19. Methenamine therapy
      20. Norepinephrine
      21. Phenobarbital
      22. Phenytoin
      23. Propoxyphene
      24. Veratrum alkaloids
  12. Any major illness in the last 3 months or any significant ongoing chronic medical illness as determined by the Investigator.
  13. Presence or history of clinically significant disorders involving cardiovascular (e.g., cardiac arrhythmias, coronary artery or organic heart disease, or hypertension), respiratory, renal, hepatic, dermatologic, musculoskeletal, gastrointestinal, immunologic, hematologic, endocrine (e.g., hyperthyroidism, hypoglycemia, or diabetes) or neurologic systems (e.g., Parkinson's disease), or psychiatric disease (e.g., depression), as determined by the Investigator.
  14. History of complaints of frequent dizziness or lightheadedness occurring more than once every week.
  15. Existence of any surgical or medical condition which, in the judgment of the Investigator, might interfere with the absorption, distribution, metabolism, or elimination of the study drug or is likely to compromise the safety of the participant.
  16. Evidence of allergy or known hypersensitivity to epinephrine, sodium metabisulfite, or to any of the components of its formulation.
  17. History or presence of difficult venipuncture for blood sampling.
  18. History or presence of open sores or areas of irritation, redness, swelling, bleeding, lesions, piercings, or mucous membranes within the mouth.
  19. Below normal serum pseudocholinesterase levels, defined as:

      a. Males i. All ages: < 5,320 U/L b. Females i. Not taking hormonal contraceptives

  <!-- -->

  1. Ages 18-39 years: < 4,260 U/L
  2. Ages > 40 years: < 5,320 U/L ii. Taking hormonal contraceptives

  <!-- -->

  1. Ages 18-41 years: < 3,650 U/L
  2. Ages > 42 years: < 5,320 U/L

  20. Any blood donation, or excess blood loss, within 30 days prior to Period 1 dosing and throughout the duration of the study. Participant agrees to continue to abstain from blood donation, outside of study activities, through end of study.

  21. Any plasma donations or plans to donate plasma within 14 days prior to Period 1 dosing and throughout the duration of the study. Participant agrees to continue to abstain from plasma donation, outside of study activities, through end of study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Cmax | 0 to 360 minutes post dose
  Maximum Epinephrine Plasma Concentration occurring at Tmax (Time to reach maximum concentration)
Tmax | 0 to 360 minutes postdose
  Time to reach maximum epinephrine plasma concentration

SECONDARY OUTCOMES:
Systolic Blood Pressure | 0 to 120 minutes postdose
  PD
Diastolic Blood Pressure | 0 to 120 minutes postdose
  PD
Pulse Rate | 0 to 120 minutes postdose
  PD

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Sweitzer, Principal Investigator — WashU Medical School
Locations (1):
- Washington University in St. Louis School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No